CLINICAL TRIAL: NCT05123079
Title: A Randomized, 3-Period Crossover Trial to Evaluate the Relative Bioavailability and Food Effect Following Single Oral Dose of Darigabat Tablet Formulations in Healthy Adult Participants
Brief Title: Relative Bioavailability and Food Effect Following Single Oral Dose of Darigabat Tablet Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVL-865-1002
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: Healthy Volunteer; Bioavailability; Food effect

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, single-center trial in healthy participants. The trial is an open-label, randomized, 3-period, 6-sequence, crossover design to investigate the relative bioavailability and effect of food of Darigabat from a single oral.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Oral Dose of 25 mg administered as 1 x 25 mg tablet, Fasted (Without Food) (Experimental): Oral Dose
  Interventions: Drug: Darigabat
- Single Oral Dose of 25 mg administered as 1 x 25 mg tablet, Fed (With food) (Experimental): Oral Dose
  Interventions: Drug: Darigabat
- Single Oral Dose of 25 mg administered as 2 x 7.5 and 2 x 5.0 mg tablets, Fasted (Without Food) (Experimental): Oral Dose
  Interventions: Drug: Darigabat

INTERVENTIONS:
Drug: Darigabat — Tablets

SUMMARY:
This is a Phase 1, single-center trial in healthy participants. This is a crossover design, open-label treatment trial with 3 periods, 6 sequences.

DETAILED DESCRIPTION:
The trial is an open-label, randomized, 3-period, 6-sequence, crossover design to investigate the relative bioavailability and effect of food on Darigabat.

ELIGIBILITY:
Inclusion Criteria:

1. Women of nonchildbearing potential and men, ages 18 to 55 years, inclusive.
2. Healthy as determined by medical evaluation by the investigator.
3. Body mass index of 18.5 to 30.0 kg/m2, inclusive, and a total body weight >50 kg (110 lbs).
4. A male participant with a pregnant or a nonpregnant partner of childbearing potential must agree to use contraception.
5. Capable of giving signed informed consent and complying with study requirements.

Exclusion Criteria:

1. Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus), malignancy (except for basal cell carcinoma of the skin and cervical carcinoma in situ, at the discretion of the investigator), hematological, immunological, neurological, or psychiatric disease.
2. Serious risk of suicide in the opinion of the investigator.
3. History of substance or alcohol-use disorder (excluding nicotine or caffeine) within 12 months prior to signing the ICF.
4. Any condition that could possibly affect drug absorption.
5. Receipt of SARS-CoV2 vaccine or booster as follows:

   * mRNA: within 14 days prior to dosing
   * Non-mRNA: within 28 days prior to dosing
6. Have recently been diagnosed with symptomatic COVID-19 or test positive for COVID-19 within 30 days prior to signing the ICF.
7. Taking any prohibited medication prior to randomization or likely to require prohibited concomitant therapy.
8. History of HIV, hepatitis B, or hepatitis C infection, or positive result for HIV, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody.
9. Positive drug screen (including nicotine and cannabinoids) or a positive test for alcohol.
10. Abnormal clinical laboratory test results or vital measurements at Screening.
11. Any other abnormal safety findings unless, based on the investigator's judgment, the findings are not medically significant and would not impact the safety of the participant or the interpretation of the trial results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Single Dose: Peak Plasma Concentrations | Day 1 to Day 4
  Peak Plasma Concentration (Cmax) for Darigabat under fasted conditions
Single Dose: Area under the plasma concentration-time curve | Day 1 to Day 4
  Area under the plasma concentration-time curve (AUC) for Darigabat under fasted conditions
Single Dose: Area under the plasma concentration-time curve from time zero to last concentration measured | Day 1 to Day 4
  Area under the plasma concentration-time curve from time zero to last concentration measured (AUClast) for Darigabat under fasted conditions
Single Dose: Time of Maximum Observed Plasma Concentrations | Day 1 to Day 4
  Time of Maximum Observed Plasma Concentrations (Tmax) for Darigabat under fasted conditions
Secondary Objective: Single Dose: Peak Plasma Concentrations | Day 1 to Day 4
  Peak Plasma Concentration (Cmax) for Darigabat under fed and fasted conditions
Secondary Objective: Single Dose: Area under the plasma concentration-time curve | Day 1 to Day 4
  Area under the plasma concentration-time curve (AUC) for Darigabat under fed and fasted conditions
Secondary Objective: Single Dose: Area under the plasma concentration-time curve from time zero to infinity | Day 1 to Day 4
  Area under the plasma concentration-time curve from time zero to infinity (AUCinf) for CVL-865 under fed and fasted conditions
Secondary Objective: Single Dose: Time of Maximum Observed Plasma Concentrations | Day 1 to Day 4
  Time of Maximum Observed Plasma Concentrations (Tmax) for Darigabat under fasted and fed conditions

SECONDARY OUTCOMES:
Secondary Outcome (AE) | Day 1 to Day 4
  Number of subjects with reported Treatment Emergent Adverse Events (TEAEs)
Secondary Outcome (ECGs) | Day 1 to Day 4
  Number of subjects with clinically significant changes in Electrocardiograms.
Secondary Outcome (Labs) | Day 1 to Day 4
  Number of subjects with clinically significant changes in laboratory measures.
Secondary Outcome (Vital Signs) | Day 1 to Day 4
  Number of subjects with clinically meaningful changes in vitals signs.
Secondary Outcome (Physical/Neurological Exam) | Day 1 to Day 4
  Number of subjects with clinically significant changes in physical and neurological exams.
Secondary Outcome (C-SSRS) | Day 1 to Day 4
  Changes from baseline of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Dandurand, MD, Study Director — Cerevel Therapeutics, LLC
Locations (1):
- Celerion Inc., Tempe, Arizona, United States